CLINICAL TRIAL: NCT04646083
Title: Depth of Maximal Insertion During Retrograde Enteroscopy Using Colonoscopy With Through-the-scope Balloon Enteroscopy (NaviAid) Compared With Using the Standard Colonoscope Alone
Brief Title: Depth of Maximal Ileal Insertion During Retrograde Enteroscopy With TTS Balloon
Acronym: NaviAid2
Status: Recruiting | Type: Observational
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Marc Zuckerman, Professor of Medicine, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: E20147
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Obscure Gastrointestinal Bleeding; Anemia, Iron Deficiency
Keywords: retrograde enteroscopy; small bowel bleeding
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Diagnostic modalities for the evaluation of small bowel pathology include video capsule endoscopy (VCE), antegrade and retrograde device-assisted enteroscopy, CT and MR enterography (1). Despite VCE being the first-line evaluation modality, it lacks interventional capability. Deep enteroscopy (DE) allows tissue sampling and other therapeutic interventions with real-time endoscopic assessment. DE is usually performed with specific endoscopes (balloon-assisted device or spiral overtube) making it time consuming and there is limited availability since special instruments and accessories are required.(1,2) The through-the-scope (TTS) balloon system consists of a balloon catheter designed for anchoring in the small bowel, inserted through the instrument channel of a standard colonoscope.(3) The catheter is advanced, the balloon is inflated and anchored in the small intestine and the endoscope slides over the guiding catheter to the inflated balloon. The most common indications for DE are obscure GI bleeding, iron deficiency anemia, abnormal capsule endoscopy and chronic diarrhea. As compared to spiral, single-or double-balloon enteroscopy, TTS (NaviAid, SMART Medical Systems Ltd, Ra'anana, Israel) is a simpler technique, which requires less investment in infrastructure. The balloon catheter is advanced blindly in front of a standard adult colonoscope as it bends around the curves of the small bowel. To prevent perforation/trauma the catheter is fitted with a soft silicone tip which easily bends under pressure.

Insertion depth can be calculated during the withdrawal of the enteroscope. The Aim of the study: To compare the depth of maximal ileal insertion between through-the-scope balloon enteroscopy (NaviAid) with enteroscopy using the adult colonoscope (Olympus CF-190) alone, in the same patient, in a prospective cohort at University Medical Center of El Paso, Texas.

DETAILED DESCRIPTION:
The Aim of the study: To compare the depth of maximal ileal insertion between through-the-scope balloon enteroscopy (NaviAid) with enteroscopy using the adult colonoscope (Olympus CF-190) alone, in the same patient, in a prospective cohort from August 1, 2020 to July 31, 2023 at University Medical Center of El Paso, Texas.

Depth of insertion is correlated with diagnostic yield, meaning that we would like to ascertain if the use of the colonoscope with NaviAid will result in greater depth of insertion and potentially more findings of small bowel abnormalities than using a colonoscope alone.

It is assumed that this is the case, but we want to show it and quantify it.

HYPOTHESIS:

The depth of ileal insertion is greater with the use of through-the-scope balloon enteroscopy (NaviAid) when compared with enteroscopy using the standard adult colonoscope (Olympus CF-190) alone.

OBJECTIVE:

To compare the depth of maximal ileal insertion between through-the-scope balloon enteroscopy (NaviAid) with the adult colonoscope (Olympus CF-190) alone, in the same patient, in a prospective cohort at University Medical Center of El Paso, Texas.

ELIGIBILITY:
Inclusion Criteria:

1. Sign Informed Consent Form
2. Patients age between 18-90 years
3. Patients in which retrograde enteroscopy is indicated for any of the following:

abnormal video capsule endoscopy non-diagnostic upper and lower endoscopy obscure gastrointestinal bleeding iron deficiency anemia non-diagnostic upper endoscopy and abnormal CT Hemodynamically stable

Exclusion Criteria:

1. Inability to sign Informed Consent Form
2. Pregnancy and breast feeding
3. Prior colon resection
4. Patients with known strictures
5. Patients with altered anatomy
6. Inadequate bowel preparation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for evaluation of obscure gastrointestinal bleeding with nondiagnostic upper and lower endoscopy with suspicion of distal small bowel source based on either abnormal videocapsule endoscopy or imaging study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
depth of maximal insertion into ileum | during the enteroscopy of the patient, about one hour
  depth of insertion is measured on withdrawal of colonoscope by estimating in 10 cm intervals

SECONDARY OUTCOMES:
diagnostic yield of retrograde enteroscopy | during the enteroscopy of the patient, bout one hour
  proportion of studies with significant findings on enterosocpy

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Zuckerman, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Science Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No